CLINICAL TRIAL: NCT05212272
Title: A Feasibility Study of Interim PET-MRI in High-grade Glioma Patients Undergoing Chemoradiation
Brief Title: MRI in High-Grade Glioma Patients Undergoing Chemoradiation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00080134; WFBCCC 91221 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2022-01-14; First posted 2022-01-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PET-MRI In High-Grade Glioma Patients Undergoing Chemoradiation (Experimental): PET scan and MRI scan of the brain, blood draw, and 1-hour of memory testing.
  Interventions: Procedure: PET-MRI Brain Scan; Diagnostic Test: Blood draw; Behavioral: Memory testing; Procedure: Optional lumbar puncture for cerebrospinal fluid collection

INTERVENTIONS:
Procedure: PET-MRI Brain Scan — Before starting radiation, participants will have a PET scan and MRI scan of the brain. After 2 to 3 weeks of radiation treatments, participants will have a repeat PET scan. Then 1 month after radiation participants will have another PET scan
Diagnostic Test: Blood draw — Blood draws will be taken at baseline, one month after radiation treatment and 3 to 4 months after radiation treatment.
Behavioral: Memory testing — 3 sessions with simple tests to evaluate how the brain is working. These tests primarily check things like memory, attention, and thought process. The whole set of tests will take 1 hour each time.
Procedure: Optional lumbar puncture for cerebrospinal fluid collection — Participants that consent for cerebrospinal fluid collection will have 6 and 20 ml of cerebrospinal collected at baseline.

SUMMARY:
The purpose of this research study is to see if investigators can predict how brain functioning changes after radiation treatment based on PET scans and blood tests. Most participants experience at least mild decreases in their memory or attention after radiation therapy. Investigators hope that PET scans, lumbar puncture, and blood tests might help investigators predict who might have larger changes in their brain function after radiation.

DETAILED DESCRIPTION:
Primary Objective: To determine the feasibility of interim PET-MRI in high-grade glioma patients undergoing chemoradiation by quantifying the proportion of high-grade glioma patients who are alive at 4 months post-radiation treatment and who have completed two PET scans and abbreviated cognitive testing pre-radiation treatment and at 4 months post radiation treatment.

Secondary Objectives

* To determine by machine learning if early changes on FDG-PET correlate with cognitive decline after radiation treatment. Cognitive impairment will be defined as a 1 standard deviation decline on any test.
* To determine if baseline serum or cerebrospinal fluid markers or the change from baseline to 1-month are associated with patients with cognitive decline at 4-months after radiation treatment (defined as a 1 standard deviation decline on any test) compared to those without decline.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of high grade glioma (grade III or IV) or WHO grade II glioma, IDH wildtype (molecular glioblastoma multiforme [GBM]).
* ≥18 years of age.
* ECOG performance status of 0 to 3
* Anticipated to receive 6 weeks of chemoradiation

Exclusion Criteria:

* Does not speak or read English
* Unable to participate in cognitive testing due to aphasia or other severe cognitive impairment as determined by the PI, or Dr. Cummings or her designee.
* Unable to give informed consent
* Past medical history of any kind of dementia or diagnosed with mild cognitive impairment prior to diagnosis with their brain tumor
* Unable to safely fast for 8 hours prior to bloodwork or 6 hours prior to PET scan
* Currently taking cognition-enhancing medications including:

  * Donepezil
  * Memantine
  * Armodafinil
  * Methylphenidate
* Pregnant or nursing mothers.
* Patients taking blood thinners will be excluded from the optional Lumbar Puncture only, they are eligible for participation in the main study-provided they meet inclusion/exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants to Complete Two PET scans | 4 months post-treatment
  Feasibility is defined as 70% of patients who complete two PET scans. This proportion and its 95% confidence interval will be calculated at 4 months
Number of Participants to Complete Cognitive Testing | 4 months post-treatment
  Using a customized abbreviated cognitive battery designed for brain tumor patients to measure a range of cognitive functions affected by cancer and radiation treatment including basic attention, information processing speed, language, learning and recent memory, executive functions (spanning verbal fluency, cognitive set-shifting, and abstract reasoning), and visual perceptual/spatial skills. Premorbid functioning (assessing cognitive reserve) will also be assessed via a single word reading test that is strongly associated with overall intellectual functioning. Most tests have multiple forms to allow for assessment at sequential time points. All tests have well-validated normative data and have been used previously with cancer patients. Fatigue, depression, anxiety, and quality of life will be evaluated simultaneously using standard and validated patient questionnaires

SECONDARY OUTCOMES:
Change in PET measure Related to Cognitive Decline after Radiation Treatment | At baseline and 4 months post-treatment
  Change in cognitive decline is defined as one standard deviation on any neurocognitive test given using the 2-sample t-test (if normally distributed; transformation may be needed) or Wilcoxon rank sum test (if not normally distributed) when appropriate. Investigators will also relate baseline PET measure and change in PET measure to the cognitive change using the Spearman's rank correlation coefficient.
Change in Cerebrospinal Fluid Biomarkers Related to Cognitive Decline after Radiation Treatment | At baseline and 4 months post-treatment
  Changes in serum and cerebrospinal fluid biomarkers will be related to the cognitive decline at 4 months using the 2-sample t-test or Wilcoxon rank sum test when appropriate. We will also relate baseline and changes in serum and CSF biomarkers to the cognitive change using the Spearman's rank correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Cramer, MD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No